CLINICAL TRIAL: NCT02168114
Title: Optical Imaging of Dystrophic and Damaged Muscle
Brief Title: Magnetic Resonance and Optical Imaging of Dystrophic and Damaged Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201602354; MD110050 (Other: Department of Defense); 536-2012 (Other: UF legacy study)
Record Dates: First submitted 2014-06-06; First posted 2014-06-20 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Exercise; Optical Imaging; Magnetic Resonance
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity | interventions — Magnetic Resonance Spectroscopy; Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duchenne Muscular Dystrophy (Experimental): This arm will only include subjects that have a confirmed diagnosis of Duchenne Muscular Dystrophy. Subjects in this arm will not undergo any exercising, and will only be imaged by Optical and Magnetic Resonance Imaging and Spectroscopy techniques at a single time point.
  Interventions: Procedure: Optical and Magnetic Resonance Imaging and Spectroscopy
- Non-affected Subjects (Experimental): This arm will contain subjects that are not affected by Duchenne Muscular Dystrophy. These subjects will undergo concentric exercising of one forearm, and eccentric exercising of the contralateral forearm. Two days following the exercising, subjects will undergo Optical Imaging and Magnetic Resonance Imaging and Spectroscopy.
  Interventions: Other: Exercising; Procedure: Optical and Magnetic Resonance Imaging and Spectroscopy

INTERVENTIONS:
Other: Exercising — This arm will only include subjects that have a confirmed diagnosis of Duchenne Muscular Dystrophy. Subjects in this arm will not undergo any exercising, and will only be imaged by Optical and Magnetic Resonance Imaging and Spectroscopy techniques at a single time point.
  Arms: Non-affected Subjects
Procedure: Optical and Magnetic Resonance Imaging and Spectroscopy — This arm will contain subjects that are not affected by Duchenne Muscular Dystrophy. These subjects will undergo concentric exercising of one forearm, and eccentric exercising of the contralateral forearm. Two days following the exercising, subjects will undergo Optical Imaging and Magnetic Resonance Imaging and Spectroscopy.

SUMMARY:
The purpose of this research study is to determine the potential of Optical Imaging techniques to detect muscle damage in boys with Duchenne Muscular Dystrophy and unaffected exercised muscle. Healthy subjects will undergo two different exercises in opposite forearms before any imaging techniques are performed. Boys with Duchenne Muscular Dystrophy will only undergo the imaging techniques without exercise.

DETAILED DESCRIPTION:
The overall objective of this proposal is to validate the potential of Optical Imaging techniques to be able to detect and quantify muscle damage in a population affected by Duchenne Muscular Dystrophy, a muscle wasting disease, and in a healthy population that has undergone temporal muscle damage resulting from an exercising intervention.

Duchenne Muscular Dystrophy is a relentlessly progressive degenerative muscle wasting disease, clinically characterized by progressive muscle weakness, a loss of ambulation, and premature mortality. Currently, no known cure exists and treatments that benefit patients diagnosed with Duchenne Muscular Dystrophy are limited. New approaches, such as cell therapy, gene transfer, and pharmacological interventions have shown promising results in animal models and human studies with great potential to develop as effective therapeutic treatments. One of the major limitations of testing these interventions; however. is the lack of effective methods to monitor cellular and tissue changes taking place in the response to therapy. The ability to determine cellular and tissue specific changes in damaged muscles in real time, non-invasively, repeatedly, without exposure to any harmful radiations, with minimal patient discomfort, and at low operating cost would enable high throughput and faster investigation of potential therapies.

The proposed study focuses on the development of Optical Imaging technologies in the near infrared range of wavelengths to differentiate damaged from normal muscle tissue. Near infrared light (700 - 900 nm) has demonstrated the ability to deeply penetrate through biological tissue, skin, and muscle without appreciable attenuation or auto-fluorescence.

The investigators anticipate that Indocyanine Green enhanced Optical Imaging can be used to image exercise induced acute muscle damage in healthy individuals and damaged muscle and in boys with Duchenne Muscular Dystrophy. It is anticipated that this work may fulfill the need for imaging biomarkers that monitor and quantify cellular damage, muscle perfusion, and drug delivery - non-invasively, using benign light, repeatedly, and in real time, with the intention of accelerating the testing of efficacy in clinical trials for neuromuscular disorders. The study is designed to determine the ability of Optical Imaging as a reliable, safe, relatively inexpensive, and facile tool to detect and quantify muscle damage. Investigators anticipate that this type of imaging modality will provide clinically useful information for diagnostic and prognostic purposes in patients with neuromuscular diseases, especially boys with Duchenne Muscular Dystrophy.

ELIGIBILITY:
Inclusion Criteria for Duchenne Muscular Dystrophy subjects:

* Diagnosis of Duchenne muscular dystrophy confirmed by 1) clinical history with features before the age of 5 years, 2) physical examination, 3) elevated serum creatine kinase level, and 4) absence of dystrophin expression as determined by immune stain or Wester blot (<2%) and/or DNA confirmation of dystrophin mutation
* Must be between 10-15 years of age.
* Must be male.

Inclusion Criteria for unaffected subjects:

* Must be older than 18 years of age.
* Must be male.

Exclusion Criteria for unaffected and Duchenne Muscular Dystrophy subjects:

* Contraindication to an Magnetic Resonance examination (e.g. aneurysm clip, severe claustrophobia, magnetic implants)
* Presence of a condition in patients that impacts muscle function or muscle metabolism (e.g. myasthenia gravis, endocrine disorder, mitochondrial disease)
* Medical condition leading to developmental delay or impaired motor control (e.g. cerebral palsy)
* Unstable medical condition (e.g. uncontrolled seizure disorder)
* Behavioral problems causing an inability to cooperate during testing
* Control subjects who are participating in sport specific training 2 times or more per week
* History of allergy to iodides

Ages: 10 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Indocyanine Green accumulation in forearm muscles | Up to 2 days
  Percentage of area with elevated Indocyanine Green in muscle will be an indicator of cell membrane damage and will be measured using Optical Imaging in the forearms of study participants.
Muscle T2 elevation in forearm muscles | Up to 2 days
  Muscle T2 is a noninvasive marker of muscle damage/inflammation and will be measured using Magnetic Resonance in the forearms of participants of this study.

SECONDARY OUTCOMES:
Delayed Onset of Muscle Soreness (DOMS) | Up to 2 days
  DOMS will be correlated to percentage of elevated pixels within forearms of study participants.
Serum Creatine Kinase | Up to 2 days
  Serum Creatine Kinase is a marker of muscle damage and will be correlated to percentage of elevated pixels within forearms of study participants

CONTACTS AND LOCATIONS:
Overall Officials: Glenn A Walter, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States